CLINICAL TRIAL: NCT03476850
Title: Quadratus Lumborum Block Versus Transversus Abdominus Plane Block for Pain Management After Donor Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Eric Bolin, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00073925
Record Dates: First submitted 2018-02-28; First posted 2018-03-26 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Kidney Donor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Prospective randomized double-blinded trial to compare TAP block versus QL block for pain management in living donor nephrectomy patients. Participants will be blinded to the type of block received and physicians will be blinded both intra- and post-op regarding which block patients received. The team who performs the block will know which block the patient received. No one else involved in the care of the patient will know. The surgery team will not know, and the primary (in the OR) anesthesia team will not know. None of the providers involved in post-operative care of the patient will know.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL Block (Active Comparator): Blocks will be performed under the supervision of a regional anesthesia attending experienced in the performance QL blocks. QL block will be performed using ropivacaine 0.375% 20ml each side for a total volume of 40cc.
  Interventions: Procedure: QL Block
- TAP Block (Active Comparator): Blocks will be performed under the supervision of a regional anesthesia attending experienced in the performance TAP blocks. TAP block will be performed using ropivacaine 0.375% 20ml each side for a total volume of 40cc.
  Interventions: Procedure: TAP Block

INTERVENTIONS:
Procedure: QL Block — Blocks will be performed under the supervision of a regional anesthesia attending experienced in the performance QL blocks. QL block will be performed using ropivacaine 0.375% 20ml each side for a total volume of 40cc.
  Arms: QL Block
Procedure: TAP Block — Blocks will be performed under the supervision of a regional anesthesia attending experienced in the performance TAP blocks. TAP block will be performed using ropivacaine 0.375% 20ml each side for a total volume of 40cc.
  Arms: TAP Block

SUMMARY:
To evaluate quadratus lumborum block effect on post operative pain scores during the first 24 hours after surgery as compared to transversus abdominis plane block after laparoscopic donor nephrectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic assisted donor nephrectomy
* Patients that have elected to have a nerve block
* 18 years of age or older
* Patients of ASA status I - III

Exclusion Criteria:

* Chronic pain or narcotic usage during the preceding 30 days
* Infection at or near the intended needle insertion site
* Complex or altered abdominal wall anatomy
* Weight <45kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QL Block | TAP Block
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QL Block | TAP Block | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.39) | 44.6 (10.4) | 45.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score
Description: NRS patient reported (number rated pain score, 0=no pain - 10=highest pain) over the first 24 hours post operative.
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
score on a scale | 5.2 (2.5) | 5.1 (2.6)
Statistical Analysis 1: Comparison: QL Block vs TAP Block; An a priori sample size calculation found 24 subjects per group (48 total) provided >80% power to detect a 2 unit difference in patient reported pain based on a 2-sided test and significance level a = 0.05 assuming at least 3 measures per subject and a within subject covariance having a compound symmetric structure with a standard deviation in pain score of 3 units and within subject correlation of 0.5; Test type: Superiority; p = .883, Mixed Models Analysis; Mean Difference (Final Values) = 0.08

2. Secondary Outcome: Total Cumulative Opioids
Description: opiate consumption first 72 hours post operatively
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents (MME)
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
morphine milligram equivalents (MME) | 74.9 (24.3) | 73.7 (32.1)
Statistical Analysis 1: Comparison: QL Block vs TAP Block; Test type: Superiority; p = .977, ANOVA; Median Difference (Final Values) = 0.25

3. Secondary Outcome: Number of Participants With Nausea or Emesis Requiring Antiemetic Medication
Description: Antiemetics given in PACU. Occurrence of nausea or emesis requiring antiemetic medication administration in PACU.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
Participants | 17 | 8
Statistical Analysis 1: Comparison: QL Block vs TAP Block; Test type: Superiority; p = .009, Chi-squared; Odds Ratio (OR) = 4.9

4. Secondary Outcome: Number of Participants With Block Related Complications
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

5. Secondary Outcome: Length of Stay in Post Anesthesia Care Unit (PACU)
Description: Duration of PACU stay.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
minutes | 79.3 (51.7) | 88.6 (31.9)
Statistical Analysis 1: Comparison: QL Block vs TAP Block; Test type: Superiority; p = .110, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 18

6. Secondary Outcome: Length of Hospital Stay
Description: The time from surgery completion to subject meeting discharge criterion.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | QL Block | TAP Block
Number analyzed (Participants) | 24 | 24
days | 1.97 (0.8) | 1.93 (0.75)
Statistical Analysis 1: Comparison: QL Block vs TAP Block; Test type: Superiority; p = .719, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.26

ADVERSE EVENTS:
Time Frame: 0-24 hours post operative
Arm/Group | QL Block | TAP Block
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03476850/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03476850/ICF_001.pdf